CLINICAL TRIAL: NCT06921044
Title: A Multicenter, Prospective Phase Ⅱ Clinical Study of R-mini-MCOP（Rituximab / Mitoxantrone Liposome / Cyclophosphamide / Vincristine / Prednisone） in the Treatment of Elderly, Previously Untreated Diffuse Large B-cell Lymphoma
Brief Title: A Study of R-mini-MCOP in the Treatment of Elderly, Previously Untreated DLBCL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xiaohui He (Other)
Collaborators: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Xiaohui He, Chief physician，Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DED-DLBCL-K15
Record Dates: First submitted 2025-02-25; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-01

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: Diffuse large B-cell lymphoma，; Mitoxantrone Hydrochloride liposomal
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Cyclophosphamide; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- R-mini-MCOP (Experimental): Rituximab ：375 mg/m2，ivgtt，d0； Mitoxantrone Liposome ： The first dose level: 6mg/m2, ivgtt, d1; The second dose level: 8mg/m2, ivgtt, d1; The third dose level: 10mg/m2, ivgtt, d1; Cyclophosphamide :400 mg/m2，ivgtt，d1； Vincristine :1mg，ivgtt，d1； Prednisone:40 mg/m2，po.，d1-5； Q3W（Every 3 Weeks）
  Interventions: Drug: R-miniMCOP:Rituximab / Mitoxantrone Liposome / Cyclophosphamide / Vincristine / Prednisone

INTERVENTIONS:
Drug: R-miniMCOP:Rituximab / Mitoxantrone Liposome / Cyclophosphamide / Vincristine / Prednisone — Rituximab ：375 mg/m2，ivgtt，d0； Mitoxantrone Liposome ： The first dose level: 6mg/m2, ivgtt, d1; The second dose level: 8mg/m2, ivgtt, d1; The third dose level: 10mg/m2, ivgtt, d1; Cyclophosphamide :400 mg/m2，ivgtt，d1； Vincristine :1mg（，ivgtt，d1； Prednisone:40 mg/m2，po.，d1-5； Q3W

SUMMARY:
Research purpose： To evaluate the efficacy and safety of R-mini-MCOP in first-line treatment of primary treatment of diffuse large B-cell lymphoma (DLBCL) in elderly patients Experimental design： Single-arm, multicenter, prospective study

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 80 years
2. The histopathological diagnosis was diffuse large B-cell lymphoma, and immunohistochemistry was positive for CD20
3. Previously untreated disease
4. Ann Arbor stage I-IV disease
5. According to Lugano2014 criteria, there must be at least one matching evaluable or measurable lesion: lymph node lesion, the length of the measurable lymph node must be greater than 1.5cm; For non-lymph node lesions, the measured extra-nodal lesions should be > 1.0cm in length;
6. ECOG score 0-4(ECOG score 0-2 after pre-treatment and before R-mini-MCOP regimen)
7. Bone marrow function: neutrophil count ≥1.5×109/L, platelet count ≥75×109/L, hemoglobin ≥80g/L (neutrophil count ≥1.0×109/L, platelet count ≥50×109/L, hemoglobin ≥75 g/L in patients with bone marrow involvement);
8. Liver and kidney function: serum creatinine ≤1.5 times the upper limit of normal value; AST and ALT ≤2.5 times the upper limit of normal (≤5 times the upper limit of normal for patients with liver invasion); Total bilirubin ≤1.5 times the upper limit of normal value (≤3 times the upper limit of normal value for patients with liver invasion;
9. Have the swallowing power
10. Life expectancy > 3 months
11. Patients fully understand the study, voluntarily participate and sign an informed consent form (ICF) -

Exclusion Criteria:

1. Previous systemic antitumor therapy (except pre-therapy used before the first cycle of R-CMOP);
2. Metastatic diffuse large B-cell lymphoma；
3. Known central nervous system lymphoma
4. Hypersensitivity to any investigational drug or its ingredients;
5. Uncontrollable systemic diseases (such as advanced infections, uncontrolled hypertension, diabetes, etc.);
6. Hepatitis B and hepatitis C active infection (hepatitis B virus surface antigen positive and hepatitis B virus DNA more than 1x103 copies /mL; More than 1x103 copies /mL of HCV RNA);
7. Human immunodeficiency virus (HIV) infection (HIV antibody positive);
8. Other serious comorbidities, intolerance to this protocol or inappropriate participation in this study (judged by the investigator)
9. Previous or current co-occurrence of other malignancies (other than non-melanoma basal cell carcinoma of the skin that is effectively controlled, breast/cervical carcinoma in situ, and other malignancies that have been effectively controlled without treatment within the past five years);
10. Inability to swallow the drug or any significant removal of the small intestine that may prevent full absorption of the drug;
11. Situations in which other investigators have determined that participation in this study is not appropriate.

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-04-16 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Complete response rate （CRR） | At the end of Cycle 2 (each cycle is 21 days)
  Complete response rate at the end of induction

SECONDARY OUTCOMES:
Overall Response (CR+PR) Rate （ORR） | At the end of Cycle 2 (each cycle is 21 days)
  Overall Response (CR+PR) rate at the end of induction
Duration of response (DOR) | From the date when criteria for response are met (CR or PR) until the date of progression or relapse. Patients without relapse or progression or death from other causes will be censored at their last assessment date (24 months from response date)
Progression-free survival (PFS) | Time between the date of enrolment and the date of disease progression, relapse or death from any cause (12,24 months)
Overall Survival (OS) | Time between the date of enrolment and the date of death from any cause (12,24, 36 and 48 months)
Event Free Survival (EFS) | From the date of enrolment to the date of disease progression, relapse from CR, initiation of subsequent systemic anti-lymphoma therapy after the least 6 cycles of RI-CHOP (each cycle is 21 days), or death whichever occurs first (24, 36 and 48 months)